CLINICAL TRIAL: NCT03535506
Title: Preoperative Palbociclib in Patients With DCIS of the Breast That Are Candidates for Surgery
Acronym: WI223281
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: lack of accrual
Sponsor: Georgetown University (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018-0075
Record Dates: First submitted 2018-03-15; First posted 2018-05-24 (Actual); Results first posted 2025-09-26 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: DCIS
Keywords: Breast Cancer; DCIS; Ductal Carcinoma In Situ; Palbociclib
MeSH Terms: conditions — Carcinoma, Intraductal, Noninfiltrating; Breast Neoplasms | interventions — palbociclib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Patients enrolled to Group A will receive a 12-day course of Palbociclib before surgery. They will receive Palbociclib 100mg PO daily x 12 days.
  Interventions: Drug: Palbociclib
- Group B (No Intervention): These patients will receive no pre-operative treatment. Core biopsies from diagnosis and material from definitive surgery will be collected for translational studies and tissue banking. They will also provide blood samples at screening and prior to definitive surgery.

INTERVENTIONS:
Drug: Palbociclib — Palbociclib capsules for oral administration contain 125 mg, 100 mg, or 75 mg of palbociclib, a kinase inhibitor.
  Other Names: Ibrance
  Arms: Group A

SUMMARY:
This is a feasibility study which will evaluate the effects of pre-operative treatment of DCIS of the breast with palbociclib. Patients with biopsy-proven DCIS are eligible for the study.

There will be 2 independent and unrelated study groups of 12 patients each, for a total of 24 patients:

1. Group A, of male or female patients treated with palbociclib single agent (n=12);
2. Group B, untreated, of male or female patients who consented translational studies in blood, as well as diagnostic and definitive surgical specimen, but not the pre-operative treatment with palbociclib (n=12).

ELIGIBILITY:
Inclusion Criteria for all patients (Groups A and B):

* Signed informed consent obtained prior to any study specific assessments and procedures
* Age ≥18 years
* Premenopausal and postmenopausal women, or men
* Current pathologic diagnosis of DCIS of the breast of any receptor status; History of previous DCIS allowed provided that the patient is currently off systemic risk-reduction endocrine therapy; History of previous invasive breast cancer adequately treated and that is currently in remission and unrelated to current DCIS (based on primary tumor location) is allowed as long as patient is currently off systemic therapy for that invasive cancer for at least 4 weeks prior to pre-treatment biopsy (diagnostic biopsy); Patients with multifocal or multicentric lesions are allowed, as long as at least one lesion is histologically confirmed DCIS and overall clinical AJCC Stage 0 or I.
* A formalin-fixed paraffin-embedded (FFPE) tumor tissue block from diagnostic biopsy must be transmitted to MedStar Georgetown University Hospital Pathology Department repository and confirmation of receipt must be available prior to enrollment.
* Positive Rb by immunohistochemistry in the DCIS component of the lesion - must be performed at CLIA-approved setting (for instance, MGUH); Rb staining will be considered positive when 1+ or above (in a scale of 0, 1+, 2+ or 3+)
* In the absence of histologic diagnosis of DCIS, patient may undergo fresh biopsy for eligibility, provided: this invasive procedure is not a Fine Needle Aspiration (FNA); AND this procedure is a core biopsy, stereotactic biopsy or incisional biopsy of the suspicious breast lesion; AND the primary lesion is not completely resected during the procedure.
* The patient is candidate for and is willing to receive definitive surgical therapy for DCIS
* ECOG performance status 0-1
* Willingness to provide a sample of tissue collected at definitive surgery for research

Inclusion criteria specific to treatment Group A:

* Patients must be able and willing to swallow and retain oral medication
* Absolute neutrophil count (ANC) ≥ 1,500/mm3
* Platelets ≥ 120,000/mm3
* Hemoglobin ≥ 10g/dL
* Total serum bilirubin ≤ ULN; or total bilirubin ≤ 3.0 × ULN with direct bilirubin within normal range in patients with documented Gilbert's Syndrome.
* Aspartate amino transferase (AST or SGOT) and alanine amino transferase (ALT or SGPT) ≤ 1.5 × institutional ULN
* Serum creatinine within normal institutional limits or creatinine clearance ≥ 50 mL/min/1.73 m2 for patients with serum creatinine levels above institutional ULN.
* Pregnancy must be ruled out: serum or urine pregnancy test must be negative within 14 days of treatment start in women of childbearing potential. Pregnancy testing does not need to be pursued in patients who are judged as postmenopausal before enrollment, or who have undergone tubal ligation, bilateral oophorectomy, total hysterectomy.
* Willingness to undergo adequate contraception if childbearing potential; women of childbearing potential and male patients randomized into treatment Group A must use adequate contraception for the duration of protocol treatment and for 3 months after the last treatment with palbociclib if they are in Group A; adequate contraception is defined as one highly effective form (i.e. abstinence, (fe)male sterilization) OR two effective forms (e.g. non-hormonal IUD and condom / occlusive cap with spermicidal foam / gel / film / cream / suppository).

Exclusion Criteria for all patients (Groups A and B):

* Concurrent therapy with other Investigational Products
* Invasive carcinoma present in the diagnostic biopsy, microinvasion is allowed
* Uncontrolled intercurrent illness including (active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, diabetes, pulmonary embolism in the past 6 months, or psychiatric illness/social situations that would limit compliance with study requirements).
* Unable to comply with study requirements
* Hormone therapies containing estrogen, progesterone, GnRH agonists and antagonists within 4 weeks from diagnostic biopsy.
* Therapy with any CDK inhibitor in the past 3 months

Exclusion criteria specific to treatment Group A:

* History of allergic reactions attributed to compounds of chemical or biologic composition similar to palbociclib
* Presence of a condition that would interfere with enteric absorption of palbociclib
* Pregnant women, or women of childbearing potential without a negative pregnancy test (serum or urine) within 7 days prior to enrollment; breastfeeding must be discontinued prior to study entry (Group A only).
* Patients on combination antiretroviral therapy, i.e. those who are HIV+ (potential for pharmacokinetic interactions or increased immunosuppression with palbociclib).
* Patients receiving any medications or substances that are potent inhibitors or inducers of CYP3A isoenzymes within 7 days of enrollment or during participation on study
* Patients with clinically significant history of liver disease, including viral or other known hepatitis, current alcohol abuse, or cirrhosis, etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2018-10-08 (Actual); Primary Completion 2023-12-06 (Actual); Study Completion 2023-12-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Candace Mainor, MD, Principal Investigator — Georgetown University
Locations (2):
- United States (2):
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Medstar Washington Hospital Center, Washington D.C., District of Columbia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Group A- Palbociclib Before Surgery: Patients enrolled to Group A will receive a 12-day course of Palbociclib before surgery. Patients will receive Palbociclib 100mg PO daily x 12 days.
- Group B- No Pre-operative Treatment: These patients will receive no pre-operative treatment. Core biopsies from diagnosis and material from definitive surgery will be collected for translational studies and tissue banking. They will also provide blood samples at screening and prior to definitive surgery.
Period: Overall Study
Arm/Group | Group A- Palbociclib Before Surgery | Group B- No Pre-operative Treatment
Started | 5 | 12
Completed | 5 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A- Palbociclib Before Surgery | Group B- No Pre-operative Treatment | Total
Number analyzed (Participants) | 5 | 12 | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 9 | 14
  >=65 years | 0 | 3 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 12 | 17
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 5 | 10 | 15
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 4 | 6
  White | 3 | 5 | 8
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Feasibility: Recruitment Rates
Description: The approach will be considered feasible if more than 50% of the enrolled patients are treated andcomplete the study.
Time Frame: 5 years
Population: Study was terminated due to lack of accural
Measure: Count of Participants; unit: Participants
Arm/Group | Group A- Palbociclib Before Surgery | Group B- No Pre-operative Treatment
Number analyzed (Participants) | 5 | 12
Participants | 5 | 11

2. Secondary Outcome: Pathologic Changes
Description: Number of patients with pathologic changes in breast tissue before and after definitive surgery.
Time Frame: 2 months
Population: Subject in group B did not have specimens collected per protocol so was not included in the analysis. Subject in Group A could not be analyzed due to no evidence of disease at the time of definitive surgery.
Measure: Count of Participants; unit: Participants
Arm/Group | Group A- Palbociclib Before Surgery | Group B- No Pre-operative Treatment
Number analyzed (Participants) | 4 | 11
Participants | 0 | 0

3. Secondary Outcome: Pathology Changes on Immunohistochemistry (IHC)
Description: Number of treated subjects with pharmacodynamic changes evaluated by IHC from diagnostic biopsy to definitive surgery.
Time Frame: 2 months
Population: Treatment arm evaluated for Changes and 1 participant had no evidence of disease at surgery so there was no surgical specimen available to evaluate.
Measure: Count of Participants; unit: Participants
Arm/Group | Group A- Palbociclib Before Surgery | Group B- No Pre-operative Treatment
Number analyzed (Participants) | 4 | 0
Participants | 4 |

4. Secondary Outcome: Toxcity Based on CTCAE
Description: Number of subjects with an adverse event reported from time of consent until up to 32 days after surgery.
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Group A- Palbociclib Before Surgery | Group B- No Pre-operative Treatment
Number analyzed (Participants) | 5 | 12
Participants | 5 | 0

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Group A- Palbociclib Before Surgery | Group B- No Pre-operative Treatment
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/12
Other Adverse Events (participants affected / at risk) | 5/5 | 0/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A- Palbociclib Before Surgery (N=5) | Group B- No Pre-operative Treatment (N=12)
Dry mouth (Gastrointestinal disorders) | 1 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal disorders - Other, specify: (Gastrointestinal disorders) | 1 (1) | 0 (0) — Dry Lips
Infections and infestations - Other, specify: (Infections and infestations) | 1 (1) | 0 (0) — Covid-19
Headache (Nervous system disorders) | 1 (2) | 0 (0)
Hallucinations (Psychiatric disorders) | 1 (1) | 0 (0)
Breast pain (Reproductive system and breast disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-01-20): https://cdn.clinicaltrials.gov/large-docs/06/NCT03535506/Prot_SAP_000.pdf